CLINICAL TRIAL: NCT02973399
Title: A Phase 1, Open-label Study of SNX-5422 Added to Ibrutinib in Chronic Lymphocytic Leukemia Subjects With Residual Disease
Brief Title: Efficacy and Safety of SNX-5422 Added to an Established Dose of Ibrutinib in CLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN1-012
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Cancer
Keywords: CLL; Leukemia, Chronic Lymphocytic; Hsp90; Ibrutinib
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — SNX-5422; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SNX-5422 plus ibrutinib (Experimental): Open-label administration of SNX-5422 capsules dosed in the morning once every other day for 21 days (11 doses) followed by a 7 day drug free period and daily with the established ibrutinib dose for 28 days of a 28-days cycle. Subjects will repeat the 28-day schedule for 2 cycles after a CR or until the cancer progresses or the subject is unable to tolerate the therapy
  Interventions: Drug: SNX-5422 plus ibrutinib

INTERVENTIONS:
Drug: SNX-5422 plus ibrutinib — SNX-5422 capsule(s) dosed every other day for 21 days out of a 28-day treatment cycle to a total dose of 56 mg/m2 SNX-5422. Subjects will self-administer daily oral ibrutinib in the afternoon at least 8 hours apart from SNX-5422 for 28 days of each cycle.
  Other Names: Imbruvica

SUMMARY:
SNX-5422 is a prodrug of SNX-2112, a potent, highly selective, small molecule inhibitor of the molecular chaperone heat shock protein 90 (HSP90). Hsp90 inhibitors may overcome ibrutinib resistance in Mantle cell lymphomas and this study will investigate whether the addition of SNX-5422 to an established dose of ibrutinib will provide clinical response in subjects who have residual disease, but have not progressed on ibrutinib after 18 months of monotherapy, and/or prevents or delays disease progression of subjects with CLL.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most prevalent leukemia in adults and is not considered curable outside of allogeneic stem cell transplantation. Significant advances have been made in the therapy, notably with the introduction of the Bruton's tyrosine kinase (BTK) inhibitor ibrutinib.

While response to ibrutinib has been high with therapy well-tolerated overall, some patients have relapsed while others have been taken off therapy for toxicity or other reasons. In addition, although remissions are durable in many patients, very few patients achieve a complete response (CR), and minimal residual disease (MRD) negativity on single agent ibrutinib has not been reported. Since it is known that for chemoimmunotherapy as well as targeted therapies such as venetoclax that attainment of a CR is associated with longer progression free survival (PFS), it is likely that deepening responses associated with ibrutinib will result in more durable remissions.

Relapse in CLL can be mediated by at least two separate mechanisms. One is by mutations in BTK, the other is through a variety of mutations in the immediate downstream target of BTK, PLCγ2. SNX-5422 is a prodrug of SNX-2112, a potent, highly selective, small molecule inhibitor of the molecular chaperone heat shock protein 90 (HSP90). Hsp90 inhibitors may overcome ibrutinib resistance in Mantle cell lymphomas and this study will investigate whether the addition of SNX-5422 to an established dose of ibrutinib will provide clinical response in subjects who have residual disease, but have not progressed on ibrutinib after 18 months of monotherapy.

Subjects will receive SNX-5422 (56 mg/m2) in the morning once every other day for 21 days (11 doses), followed by a 7-day drug-free period. Subjects will continue to receive daily oral ibrutinib at their established dose level in the afternoon

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older
* A diagnosis of CLL as defined by IWCLL 2008 criteria and currently on treatment with ibrutinib for at least 18 months with residual disease and without evidence of disease progression.
* No more than 4 prior lines of anti leukemia therapy (not including ibrutinib)
* Life expectancy of at least 9 months
* Karnofsky performance score 70
* Adequate baseline laboratory assessments
* Signed informed consent form
* Recovered from toxicities of previous anticancer therapy to CTCAE Grade ≤ 1
* Subjects with reproductive capability must agree to practice adequate contraception methods.

Exclusion Criteria:

* Subjects experiencing toxicity with ibrutinib
* Prior treatment with any Hsp90 inhibitor.
* Major surgery or significant traumatic injury within 4 weeks of starting study treatment.
* Conventional chemotherapy or radiation within 4 weeks.
* The need for treatment with medications with clinically-relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422
* Screening ECG QTc interval 470 msec for females, 450 msec for males.
* At increased risk for developing prolonged QT interval unless corrected to within normal limits prior to first dose of SNX-5422
* Patients with chronic diarrhea or with Grade 2 or greater diarrhea despite appropriate medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption or could alter the assessment of safety
* History of documented adrenal dysfunction not due to malignancy.
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Use of an investigational treatment (except for ibrutinib) from 30 days prior to the first dose
* Glaucoma, retinitis pigmentosa, macular degeneration, or any retinal changes detected by ophthalmological examination that are considered clinically important by examiner.
* Psychological or social reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of the combination of SNX-5422 and ibrutinib | 6 months
  Proportion of subjects obtaining a complete response at the end of 6 SNX-5422 treatment cycles

SECONDARY OUTCOMES:
Number of subjects reporting adverse events | Day 28 of each 4 week cycle from randomization up to 52 weeks
  Frequency and severity of adverse events
Complete response at 12 months | 12 months
  Proportion of subjects obtaining a complete response at the end of 6 SNX-5422 treatment cycles
Improved Clinical Status | 6 months
  Proportion of subjects obtaining improvement in clinical status (i.e., Stable Disease becoming Partial Response) at the end of 6 SNX-5422 treatment cycles
Progression free survival of patients receiving ibrutinib plus SNX-5422 | Up to 52 weeks
  Elapsed time for each subject from randomization to continued survival up to 52 weeks

OTHER OUTCOMES:
BTK Mutation Level | 6 and 12 months
  Change from baseline in percent of CLL cells with Bruton's Tyrosine Kinase mutations at the end of 6 and 12 treatment cycles

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Wexner Medical Center, Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No